CLINICAL TRIAL: NCT04190459
Title: Quality of Life 10 Years After Bariatric Surgery
Acronym: Qol-10
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Stefura, Reasearch Associate, PhD student at 2nd Department of General Surgery, Principal Investigator, Medical Doctor, Jagiellonian University
Other Study IDs: KBET/156/B/201
Record Dates: First submitted 2019-11-27; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSG: laparoscopic sleeve gastrectomy
  Interventions: Procedure: LSG
- LRYGB: laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: LRYGB

INTERVENTIONS:
Procedure: LSG — Bariatric surgery
  Groups: LSG
Procedure: LRYGB — Bariatric surgery
  Groups: LRYGB

SUMMARY:
Importance: Improvement of the QoL after bariatric surgery is an important outcome of the treatment. The investigators believe that assessment of distant QoL results, could provide new insight into effectiveness of most popular bariatric procedures.

Objective: The investigators aim to analyze the bariatric surgery effect on the long term QoL, considering the type of surgery.

Design: A cohort study including patients undergoing bariatric surgery. Setting: One academic referral center. Exposures: Patients undergo Laparoscopic Sleeve Gastrectomy or Laparoscopic Roux-en-Y Gastric Bypass . Surgical technique is standardized and consistent in the whole study group.

Main Outcomes and Measures: The main outcome is the change of QoL after bariatric surgery. It is assessed in three different time points: pre-surgery, first follow up (1 year after surgery) and second follow-up (10 years after surgery). The investigators use two licensed and standardized questionnaires: (Short Form Health Survey) and MA-QoLQII (Moorehead-Ardelt Quality of Life Questionnaire II).

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study
* meeting the eligibility criteria for bariatric treatment, either for laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (LRYGB).

Exclusion Criteria:

* previous bariatric procedures

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Initially the investigators included 65 patients undergoing surgical treatment for morbid obesity [39 females (60%) and 26 males (40%)]. Mean age was 42.75 years. Overall, 34 patients underwent LSG (52.3%) and 31 patients underwent LRYGB (47.7%). Mean initial body weight was 146.2 kg, mean BMI before surgery was 50.44 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Quality of life measured as a Short Form Health Survey - 36 score. | 10 years
  To assess the quality of life of included patients the investigators used licensed and standardized questionnaire, which is designed for medical purposes: SF-36 (Short Form Health Survey). It is scale with minimal value being 0 and maximal value being 100 scale. Higher score means better outcome.
Quality of life measured as a Moorehead-Ardelt Quality of Life Questionnaire II score. | 10 years
  To assess the quality of life of included patients the investigators used licensed and standardized questionnaire, which is designed for medical purposes: MA-QoLQII (Moorehead-Ardelt Quality of Life Questionnaire II). The MA-QoLQII questionnaire has six dimensions. The MA II questionnaire is used as a part of the Bariatric Analysis and Reporting Outcome System (BAROS) and assesses the patients subjective impression of quality of life in the areas of general self-esteem, physical activity, social contacts, satisfaction concerning work, pleasure related to sexuality and focus on eating behavior. Each item is scored from-0.5 to +0.5. The total score consists of the sum of the six dimensions with a range of -3 to +3. A total score of 1.1 to 2 is considered "good", above 2.1 is"very good".

SECONDARY OUTCOMES:
Weight change | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No